CLINICAL TRIAL: NCT05726903
Title: Counseling Among Gender Diverse Adolescents Who Use Depot Medroxyprogesterone
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 22-1037
Record Dates: First submitted 2023-01-11; First posted 2023-02-14 (Actual); Results first posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Gender Dysphoria, Adolescent
MeSH Terms: conditions — Gender Dysphoria | interventions — DEPO; N,N-dimethyl-4-anisidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Depo SC Home (Experimental): Participants will be given instructions on home administration of DMPA SC and be provided with all necessary supplies.
  Interventions: Drug: Depo-subQ Provera Injectable Product

INTERVENTIONS:
Drug: Depo-subQ Provera Injectable Product — SC Injection at Home
  Other Names: Depo, DMPA

SUMMARY:
Recommendations regarding contraceptive counseling and reproductive health differ amongst transgender and gender diverse (TGD) youth compared to cis-gender youth. Limited existing literature demonstrates the need for contraceptive counseling that moves beyond cis- and heteronormative assumptions that start with pregnancy prevention and address concerns at the intersection of gender identity.

The Investigator's qualitative study will focus on creating best practices regarding equitable contraceptive counseling for TGD youth. The Investigator will recruit transgender youth who are assigned female at birth, and currently or interested in using depo medroxyprogesterone (DMPA). Through focus groups and semi-structured interviews, the investigator hopes to guide providers in creating best practices and more equitable contraceptive counseling for TGD youth and measure satisfaction of DMPA in TGD youth.

DETAILED DESCRIPTION:
Recommendations regarding contraceptive counseling and reproductive health differ amongst transgender and gender diverse (TGD) youth compared to cis-gender youth. TGD youth face unique health disparities including increased risk of sexually transmitted infections, sexual abuse and violence, and unwanted pregnancies. TGD youth also face inequities within the healthcare system including lack of access to providers and delay or avoidance of care. Both patients and providers also have misconceptions around pregnancy risk in transgender individuals assigned female at birth (AFAB) who are sexually active with people assigned male at birth. Limited existing literature demonstrates the need for contraceptive counseling that moves beyond cis- and heteronormative assumptions that start with pregnancy prevention and address concerns at the intersection of gender identity.

The Investigator's qualitative study will focus on creating best practices regarding equitable contraceptive counseling for TGD youth. The Investigator will recruit transgender youth who are AFAB, and currently or interested in using depo medroxyprogesterone (DMPA). Through focus groups and semi-structured interviews, the investigator hopes to gain the perspectives of and experiences of TGD youth with self-and clinic- administered DMPA. The investigator hopes the results of this study can guide providers in creating best practices and more equitable contraceptive counseling and measure to satisfaction of DMPA for TGD youth.

ELIGIBILITY:
Inclusion Criteria:

* between the ages of 15-21,
* currently receiving care at one of the clinic sites, assigned female at birth, identify as transgender or gender diverse , and are currently using or are interested in using DMPA.

Exclusion Criteria:

* Any contraindications to DMPA (based on any category 3 or 4 recommendations from the CDC MEC guidelines)

Ages: 15 Years to 21 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Assigned female at birth. Gender identity, transgender or gender diverse. Our qualitative study will focus on creating best practices regarding equitable contraceptive counseling for transgender and gender diverse youth.
Enrollment: 35 (Actual)
Dates: Start 2022-12-06 (Actual); Primary Completion 2023-11-17 (Actual); Study Completion 2023-11-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eva M Dindinger, MPH, Study Chair — University of Colorado, Denver
Locations (1):
- Comprehensive Women's Health Center, Denver, Colorado, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Depo SC Home
Started | 35
Completed | 21
Not Completed | 14

BASELINE CHARACTERISTICS:
Arm/Group | Depo SC Home
Number analyzed (Participants) | 35
Age, Categorical [Count of Participants; unit: Participants] — Population: Missing data for 1 person
  Participants
    number analyzed (Participants) | 34
    <=18 years | 17
    Between 18 and 65 years | 17
    >=65 years | 0
Age, Continuous [Median (Full Range); unit: years] | 17.5 [15 to 21]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 29
  More than one race | 5
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 35

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Satisfied With Self-Administered DMPA at Initiation
Description: Patient satisfaction with DMPA as assessed by thematic analysis of audio-recorded focus groups of each individual participant. Satisfaction will be measured through thematic analysis as the transcripts for the focus groups are coded, identifying phrases and words relating to satisfaction or dissatisfaction with their injection experience. Focus groups will be led by a member of the trans-masculine young adult community who will be trained on focus group procedures. Guides will be developed from a collaboration between experts in gender-affirming care.
Time Frame: within 6 months of first DMPA administration
Measure: Count of Participants; unit: Participants
Groups:
- DMPA SC Users: Participants will be given instructions on home administration of DMPA SC and be provided with all necessary supplies.
  Depo-subQ Provera Injectable Product: SC Injection at Home
Arm/Group | DMPA SC Users
Number analyzed (Participants) | 17
Participants | 17

2. Primary Outcome: Number of Participants Satisfied With DMPA in an Office Setting
Description: Patient satisfaction with DMPA as assessed by thematic analysis of audio-recorded focus groups of each individual participant. Satisfaction will be measured through thematic analysis as the transcripts for the focus groups are coded, identifying phrases and words relating to satisfaction or dissatisfaction with their injection experience. Focus groups will be led by a member of the trans-masculine young adult community who will be trained on focus group procedures. Guides will be developed from a collaboration between experts in gender-affirming care.
  Patients who elect for DMPA administration in an office setting will not undergo individual interviews.
Time Frame: within 2 months of first DMPA administration
Measure: Count of Participants; unit: Participants
Groups:
- Depo Office: Patient received routine Depo Provera in the office
Arm/Group | Depo Office
Number analyzed (Participants) | 4
Participants | 4

ADVERSE EVENTS:
Time Frame: Adverse event data was collected through the end of the study (approximately 1 year after initial participant enrolled).
Arm/Group | Depo SC Home
All-Cause Mortality (participants affected / at risk) | 0/35
Serious Adverse Events (participants affected / at risk) | 0/35
Other Adverse Events (participants affected / at risk) | 0/35

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-09-16): https://cdn.clinicaltrials.gov/large-docs/03/NCT05726903/Prot_SAP_000.pdf